CLINICAL TRIAL: NCT02813824
Title: Assessment of the Effect of a Daily Chemoprevention by Low-dose Aspirin of New or Recurrent Colorectal Adenomas in Patients With Lynch Syndrome
Brief Title: Effect of Chemoprevention by Low-dose Aspirin of New or Recurrent Colorectal Adenomas in Patients With Lynch Syndrome
Acronym: AAS-Lynch
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P130937
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — acetylsalicylic acid lysinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aspirin300 (Active Comparator): Acetylsalicylic acid 300 mg tablet by mouth, daily dose during 4 years
  Interventions: Drug: Acetylsalicylic acid lysinate 300 mg
- Placebo300 (Placebo Comparator): Placebo (like Acetylsalicylic acid 300 mg) tablet by mouth, daily dose during 4 years
  Interventions: Drug: Placebo (for Aspirin 300)
- Aspirin100 (Active Comparator): Acetylsalicylic acid 100 mg tablet by mouth, daily dose during 4 years
  Interventions: Drug: Acetylsalicylic acid lysinate 100 mg
- Placebo100 (Placebo Comparator): Placebo (like Acetylsalicylic acid 100 mg) tablet by mouth, daily dose during 4 years
  Interventions: Drug: Placebo 100 (for Aspirin 100)

INTERVENTIONS:
Drug: Acetylsalicylic acid lysinate 300 mg — Daily dose during 4 years
  Other Names: Aspirin300
  Arms: Aspirin300
Drug: Placebo (for Aspirin 300) — Daily dose during 4 years
  Other Names: Placebo300
  Arms: Placebo300
Drug: Acetylsalicylic acid lysinate 100 mg — Daily dose during 4 years
  Other Names: Aspirin100
  Arms: Aspirin100
Drug: Placebo 100 (for Aspirin 100) — Daily dose during 4 years
  Other Names: Placebo100
  Arms: Placebo100

SUMMARY:
The proposed trial will evaluate the effect of aspirin 300 mg/d and 100 mg/d during 4 years vs placebo, in a 4 groups randomised parallel design in Lynch syndrome patients: patients with proven carriers of pathological mutations in mismatch repairs genes and patients with personal and family history characterizing Lynch syndrome according to modified Amsterdam criteria without proven mutation, aged more than 18 years with signed informed consent. The main hypothesis to be tested is that aspirin could decrease colorectal adenoma recurrence evaluated during high quality follow-up by colonic chromo-endoscopy in Lynch syndrome patients. The trial will also explore: (i) colorectal neoplasia recurrence according to different germline alteration in mismatch repair genes, (ii) observance to chemoprevention in Lynch syndrome patients, (iii) the burden of adverse events attributable to aspirin in Lynch syndrome patients, (iv) the dose-effect of aspirin on adenomatous polyp burden. All pathological samples will be reviewed using a centralized procedure. The INCA regional network organization and the HNPCC patient organization will allow the recruitment and the follow-up of a large number of patients with well characterised Lynch syndrome.

DETAILED DESCRIPTION:
Lynch syndrome (LS) is the most common inherited colorectal cancer syndrome, and results from germline mutations in mismatch repair genes that confer a high lifetime risk of colorectal cancer (CRC) (60 to 70%). Most CRCs arise from asymptomatic polyps. Development of such polyps into cancer can be prevented if polyps are detected early by endoscopy and removed. Colonoscopy is proposed every 2 years in LS patients more than 25 years old, and every year when colonic neoplasia has been detected. Efficient chemoprevention has the potential to represent a cost-effective intervention in these patients and could allow a delay in colonoscopic surveillance.

Several epidemiological studies have shown that regular use of low dose aspirin (75 to 300 mg/d) is associated with a 20 to 30 % reduction in the risk of sporadic colonic polyps and CRC. Four randomised controlled trials (RCT) have also shown a decrease in colorectal polyp recurrence. In a pooled analysis of cardio-vascular prevention RCTs, as well as in a meta-analysis, daily aspirin was associated with a reduced risk of CRC and CRC associated mortality. Aspirin preventive benefit is expected to outweigh its putative side effects in high risk patients. The CAPP2 study in Lynch syndrome patients showed that aspirin (300 mg x2/d) did not reduce significantly the risk of colorectal neoplasia after 29 months, but an extended follow-up (mean 56 months) showed a reduction in colorectal cancer in the aspirin group. In this study, the endoscopic follow-up was not optimal with a relatively low detection rate of colorectal neoplasia according to usual reported rate when chromo-endoscopy is performed. So, the real effect and clinical benefit of aspirin are still to be characterised in Lynch syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Lynch syndrome bearing an alteration of "mismatch repair" genes or,when no characteristic alteration has been found, with a personal or family history of Lynch syndrome according to modified Amsterdam criteria
* Aged more than 25 years, et aged more than 18 years with an early familial history and any reason to perform a colonoscopy every 2 years
* Aged less than 75 years

Exclusion Criteria:

* Known allergy to aspirin (including a history of asthma induced by the administration of salicylates or substances with similar activity, including non-steroidal anti-inflammatory)
* Need for a prolonged treatment (prevention of cardio-vascular risk) or repeated treatments (recurring migraines) using aspirin or another non-steroidal anti-inflammatory drug (NSAID)
* Pregnancy or breast feeding
* Participation to another clinical trial during the 12 weeks before inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients with at least one adenoma seen on chromo-endoscopy 48 months after complete withdrawal of polyps and initiation of treatment (aspirin or placebo) | 4 years
  To look for a preventive effect of low-dose aspirin (100 or 300 mg/d) compared with placebo on new or recurrent colorectal adenomas in patients with Lynch syndrome

SECONDARY OUTCOMES:
Delay between the onset of 1 adenoma after complete resection of polyps and date of start of treatment (aspirin vs placebo) | 24 and 48 months
Number of patients who presented an adenoma during follow-up based on the gene reached (MLH1, MSH2, MSH6, PMS2, or without other identified anomalies) | 24 and 48 months
Load serrated polyps after 24 and 48 months of treatment | 24 and 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert BENAMOUZIG, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soualy A, Deutsch D, Benallaoua M, Ait-Omar A, Mary F, Helfen S, Boubaya M, Levy V, Benamouzig R; AAS-Lynch group. Effect of chemoprevention by low-dose aspirin of new or recurrent colorectal adenomas in patients with Lynch syndrome (AAS-Lynch): study protocol for a multicenter, double-blind, placebo-controlled randomized controlled trial. Trials. 2020 Sep 4;21(1):764. doi: 10.1186/s13063-020-04674-8. PMID 32887653